CLINICAL TRIAL: NCT05327205
Title: Chest and Abdominal Compression Versus PROne Position
Acronym: CA_C_PRO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CA_C_PRO
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a severe pulmonary insult responsible for major, life-threatening hypoxemia. The alteration of hematosis is secondary to alveolar edema, following damage to the alveolocapillary barrier in response to a systemic inflammatory process. The presence of fluid effusion within the alveolar sacs and the modification of type II pneumocyte activity due to the presence of numerous pro-inflammatory mediators will lead to a quantitative and qualitative alteration of the surfactant. At the same time, leukocyte infiltration will lead to an alteration of the support tissue and to the accumulation of cellular debris. All these elements will lead to a heterogeneous loss of aeration of the lung. In addition, the alveolar units are compressed by the entire lung parenchyma due to the effect of gravity on the edematous tissue.

The treatment of ARDS is based on the antagonistic need to maintain hematosis and reduce parenchymal insult secondary to mechanical ventilation. Optimization of mechanical ventilation consists in reducing the volume of gas administered at each respiratory cycle and in limiting thoracic parietal stress by the use of curares. More recently, the interest of the ventral decubitus position has been demonstrated. During such a maneuver, the posterior pulmonary parenchymatous zones, usually subjected to gravity in the supine position, will be able to re-expand under the effect of the prone position and of the positive pressure induced by the ventilator. The increase in parietal elastance, due to the compression of the thorax between the posterior part of the trunk and the bed, also contributes to an improvement in the distribution of inhaled gases within the pulmonary parenchyma by limiting the loss of energy, transmitted directly to the wall. The ventral decubitus position allows to redistribute the ventilation in territories which were not aired before but which participate to the respiratory exchanges because they are still perfused and thus to improve the pulmonary compliance measured.

Although described as an atypical form, SARS-CoV-2 infection can lead to ARDS with severe forms of viral pneumonia and thus require prone positioning.

While this results in improved oxygenation and compliance, prone positioning is accompanied by a risk of complications such as pressure sores, described as the most frequent. In addition, the massive influx of patients and more generally the lack of personnel during pandemic peaks has made the application of prone position sometimes complex because it requires human resources. As a result, the benefit/risk ratio of the maneuver is difficult to determine because not all patients respond in the same way to prone positioning. It appeared essential to be able to predict the expected benefit of the prone position before performing the procubitus maneuver.

The application of thoracic and abdominal pressures, as part of the respiratory management of patients, is a technique commonly used by physiotherapists. Investigators have demonstrated a similar change in measured lung parenchymal compliance during manual compression of a patient's chest and during prone positioning. In the context of the epidemic, investigators used this test systematically to determine which patients were most likely to benefit from prone positioning and for whom the available resources should be concentrated at any given time.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient hospitalized in the ICU for acute respiratory distress syndrome at Covid-19
* Ventilated intubated patient for whom prone sessions were offered
* Patient who received respiratory physical therapy sessions on the same day as the prone position
* French-speaking patient

Exclusion Criteria:

* Non-intubated patient performing vigorous prone sessions
* Patient on invasive mechanical ventilation for another etiology than Covid-19
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were admitted to the ICU for acute respiratory distress syndrome at COVID-19 between 04/10/2021 and 04/01/2022.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of thoracic compression on motor pressure | Day 1
  This outcome corresponds to the motor pressure measured during inspiration (in cmH2O) under two specific conditions: during manual pressure and during prone position.

SECONDARY OUTCOMES:
Response to thoracic and/or abdominal pressure and prone position on resistive pressure | Day 1
  This outcome corresponds to the resistive pressure measured at inspiration (in cmH2O) during manual pressure and during prone position.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Romanet, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Gattinoni L, Taccone P, Carlesso E, Marini JJ. Prone position in acute respiratory distress syndrome. Rationale, indications, and limits. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1286-93. doi: 10.1164/rccm.201308-1532CI. PMID 24134414
- [Background] Villar J. What is the acute respiratory distress syndrome? Respir Care. 2011 Oct;56(10):1539-45. doi: 10.4187/respcare.01395. PMID 22008395
- [Background] Fan E, Brodie D, Slutsky AS. Acute Respiratory Distress Syndrome: Advances in Diagnosis and Treatment. JAMA. 2018 Feb 20;319(7):698-710. doi: 10.1001/jama.2017.21907. PMID 29466596
- [Background] Munshi L, Del Sorbo L, Adhikari NKJ, Hodgson CL, Wunsch H, Meade MO, Uleryk E, Mancebo J, Pesenti A, Ranieri VM, Fan E. Prone Position for Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S280-S288. doi: 10.1513/AnnalsATS.201704-343OT. PMID 29068269
- [Background] Tirolien JA, Garnier M. [COVID-19, an atypical acute respiratory distress syndrome]. Prat Anesth Reanim. 2020 Sep;24(4):225-229. doi: 10.1016/j.pratan.2020.07.001. Epub 2020 Jul 10. French. PMID 32837209
- [Background] Borges LF, Saraiva MS, Saraiva MAS, Macagnan FE, Kessler A. Expiratory rib cage compression in mechanically ventilated adults: systematic review with meta-analysis. Rev Bras Ter Intensiva. 2017 Jan-Mar;29(1):96-104. doi: 10.5935/0103-507X.20170014. PMID 28444078
- [Background] Sweeney RM, McAuley DF. Acute respiratory distress syndrome. Lancet. 2016 Nov 12;388(10058):2416-2430. doi: 10.1016/S0140-6736(16)00578-X. Epub 2016 Apr 28. PMID 27133972